CLINICAL TRIAL: NCT06633666
Title: Acupuncture for Long COVID Neuropsychiatric Symptoms: a Pragmatic,Randomized Clinical Trial
Brief Title: Acupuncture for Post COVID-19 Condition (Long COVID) Neuropsychiatric Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Visiting Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023Cmdevfund
Record Dates: First submitted 2024-10-05; First posted 2024-10-09 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Long Covid19; Neuropsychiatric Symptom; Acupuncture
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participants will be assigned to the treatment group or the control group according to the ratio of 1:1. This process is carried out by an independent researcher (Research Assistant), and the evaluators and outcome assessor will not know the grouping of the participants until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The acupuncture intervention will be conducted for 2 sessions per week during a 12-week treatment duration and will be followed up at week 18. This research is based on the TCM theory of individualized acupuncture. Qualified participants will first conduct TCM syndrome differentiation according to the five main manifestations of Long COVID neuropsychiatric symptoms including fatigue, anxiety/depression, cognitive impairment, memory loss, and insomnia. They will be divided into four treatment groups according to their main clinical symptoms, and the participants in the treatment group will be treated with the selected acupoints according to their disease category.
  The selection of the acupoints for each syndrome type are formulated with reference to the 13th Five-Year Plan Textbook "Acupuncture and Moxibustion Therapy" published by the China Press of Traditional Chinese Medicine Co.,Ltd.
  Interventions: Device: Acupuncture
- Conventional treatment (No Intervention): The control group will not receive acupuncture therapy. This study does not require the use of a placebo.

INTERVENTIONS:
Device: Acupuncture — 1. Fatigue Principal points: Pishu (BL 20), Ganshu (BL 18), Shenshu (BL 23), Baihui (GV 20), Guanyuan (RN 4), Zusanli (ST 36), Sanyinjiao (SP 6)
  2. Anxiety/ depression Principal points: Yintang (EX-HN3), Baihui (GV 20), Taichong (LR 3), Neiguan (PC 6), Danzhong (RN 7)
  3. Cognitive impairment/ memory loss Principal points: Baihui (GV 20), Sishencong (EX-HN1), Fengfu (GV 16), Taixi (K 13), Xuanzhong (GB 39), Zusanli (ST 36)
  4. Insomnia Principal points: Zhaohai (K 16), Shenmai (BL 62), Shenmen (HT 7), Sanyinjiao (SP 6), Anmian (EX-HN22), Sishencong (EX-HN1)
  Arms: Acupuncture

SUMMARY:
In this study, a 12-week pragmatic, randomized, double-blinded clinical trial will be conducted to evaluate the efficacy of acupuncture for the treatment of long Covid neuropsychiatric symptoms and provide reference for clinical non-drug treatment.

DETAILED DESCRIPTION:
This is a pragmatic, randomized, double-blinded clinical trial on acupuncture for treating neuropsychiatric symptoms in long Covid patients. A total of 160 participants will be diagnosed by a registered Chinese medicine practitioner and randomly assigned to the acupuncture and the control group with a 1:1 ratio. The acupuncture group will receive 24 sessions of interventions during a 12-week treatment duration (2 sessions per week) and will be followed up at week 18. The control group will only receive conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* meet the clinical diagnosis of Long COVID by the World Health Organization (WHO), with no neuropsychiatric symptoms 1 year before infection with Covid-19, and continue to have at least one neuropsychiatric symptom for 2 months after SARS-CoV-2 turned negative 3 months above;
* aged 12 to 80 years;
* willing and able to consent, and complete all assessment and study procedures

Exclusion Criteria:

* patients with a history of chronic neuropsychiatric symptoms;
* cardiovascular diseases pre-existing to the Covid-19 episode such as arrhythmia, heart failure, myocardial infarction, and patients with cardiac pacemakers;
* documented pre-existing history of psychiatric illness, including substance abuse;
* suicidal tendencies (attempted suicide in the 12 months before the study);
* any chronic or remote neurological disorder (i.e. stroke, head trauma, epilepsy, tumor);
* those who participated in other clinical trials within one month;
* pregnant or lactating female patients;
* have surgery within two months before the study or will have a scheduled surgery during the study;
* acute brain injury or acute encephalopathy from another etiology than Covid-19 (e.g., sepsis, liver or renal failure, alcohol or drug withdrawal, drug toxicity);
* open-heart cardiac surgery or cardiac arrest during the last 6 months;
* patients who received acupuncture treatment 1 month before the start of the study;
* patients who were unable to complete the assessment during screening due to severe mental, cognitive, or emotional impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive score on the Chinese version of the Mini-Mental State Examination (MMSE) scale | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  The MMSE can evaluate of five different domains of cognitive functions: (1) Orientation, with a maximum of 10 points, (2) Memory, with a maximum of 6 points, (3) Attention and calculation, with a maximum of 5 points, (4) Language, with a maximum of 8 points, and (5) Design copying, with a maximum of 1 point. It has a maximum score of 30, with MMSE score denotes severity of cognitive impairment as follows; mild: MMSE 21 to 24, moderate: MMSE 10 to 20, severe: MMSE less than 10.

SECONDARY OUTCOMES:
Depression on the Chinese Beck Depression Inventory (CBDI) | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  The scale has a total of 21 questions, with an overall score of 63, 14-19 being mild depression, 20-28 being moderate depression, and above 29 being severe depression.
Score of Insomnia Severity Index (ISI) | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  The Insomnia Severity Index in Chinese includes 5 questions to assess the severity and impact of insomnia, on an 0 to 4 scale, with the higher score reflecting worse insomnia symptoms.
Score of Brief Fatigue Inventory-Taiwanese (BFI-T) Form | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  BFI-T form is to assess the severity of fatigue and the impact of fatigue on daily functioning. Scoring Respondents rate each item on a 0-10 numeric scale, with 0 meaning "no fatigue" and 10 meaning "fatigue as bad as you can imagine." Scores are categorized as Mild (1-3), Moderate (4-6), and Severe (7-10).
Hamilton Depression Scale (HAMD) | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  A validated 24-item scale used to assess depressive severity across emotional, cognitive, and somatic domains. Scores range as follows: 0-7 (normal), 8-17 (mild depression), 18-24 (moderate depression), and ≥25 (severe depression), with higher scores indicating more severe depressive symptoms.
Hamilton Anxiety Rating Scale (HAMA) | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  A 14-item scale for assessing anxiety symptoms across somatic and psychological domains. Scoring ranges are: 0-7 (normal), 8-14 (mild anxiety), 15-28 (moderate anxiety), and ≥29 (severe anxiety), with higher scores indicating greater anxiety severity.
Traditional Chinese Medicine Symptom Scale | At baseline (before intervention), at 6, 12 weeks (the end of intervention), at 18 weeks (follow-up)
  A TCM-specific symptom scale following "Guidelines for Clinical Research on New Chinese Medicine," assessing syndrome severity based on TCM diagnostics. Scores quantify symptom burden with defined thresholds for mild, moderate, and severe syndrome levels, enabling standardized assessment of TCM syndrome differentiation.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jue Wei, MD., Study Chair — Hong Kong Baptist University
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

REFERENCES:
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Taquet M, Dercon Q, Luciano S, Geddes JR, Husain M, Harrison PJ. Incidence, co-occurrence, and evolution of long-COVID features: A 6-month retrospective cohort study of 273,618 survivors of COVID-19. PLoS Med. 2021 Sep 28;18(9):e1003773. doi: 10.1371/journal.pmed.1003773. eCollection 2021 Sep. PMID 34582441
- [Background] Suzuki M, Yokoyama Y, Yamazaki H. Research into acupuncture for respiratory disease in Japan: a systematic review. Acupunct Med. 2009 Jun;27(2):54-60. doi: 10.1136/aim.2009.000471. PMID 19502460
- [Background] von Trott P, Oei SL, Ramsenthaler C. Acupuncture for Breathlessness in Advanced Diseases: A Systematic Review and Meta-analysis. J Pain Symptom Manage. 2020 Feb;59(2):327-338.e3. doi: 10.1016/j.jpainsymman.2019.09.007. Epub 2019 Sep 18. PMID 31539602
- [Background] Cheong KB, Zhang JP, Huang Y, Zhang ZJ. The effectiveness of acupuncture in prevention and treatment of postoperative nausea and vomiting--a systematic review and meta-analysis. PLoS One. 2013 Dec 13;8(12):e82474. doi: 10.1371/journal.pone.0082474. eCollection 2013. PMID 24349293
- [Background] Zhang Y, Lin L, Li H, Hu Y, Tian L. Effects of acupuncture on cancer-related fatigue: a meta-analysis. Support Care Cancer. 2018 Feb;26(2):415-425. doi: 10.1007/s00520-017-3955-6. Epub 2017 Nov 11. PMID 29128952
- [Background] Lee SH, Lim SM. Acupuncture for insomnia after stroke: a systematic review and meta-analysis. BMC Complement Altern Med. 2016 Jul 19;16:228. doi: 10.1186/s12906-016-1220-z. PMID 27430619
- [Background] Amorim D, Amado J, Brito I, Fiuza SM, Amorim N, Costeira C, Machado J. Acupuncture and electroacupuncture for anxiety disorders: A systematic review of the clinical research. Complement Ther Clin Pract. 2018 May;31:31-37. doi: 10.1016/j.ctcp.2018.01.008. Epub 2018 Jan 31. PMID 29705474
- [Background] Flower A, Witt C, Liu JP, Ulrich-Merzenich G, Yu H, Lewith G. Guidelines for randomised controlled trials investigating Chinese herbal medicine. J Ethnopharmacol. 2012 Apr 10;140(3):550-4. doi: 10.1016/j.jep.2011.12.017. Epub 2011 Dec 23. PMID 22210103
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Kahn RS, Fleischhacker WW, Boter H, Davidson M, Vergouwe Y, Keet IP, Gheorghe MD, Rybakowski JK, Galderisi S, Libiger J, Hummer M, Dollfus S, Lopez-Ibor JJ, Hranov LG, Gaebel W, Peuskens J, Lindefors N, Riecher-Rossler A, Grobbee DE; EUFEST study group. Effectiveness of antipsychotic drugs in first-episode schizophrenia and schizophreniform disorder: an open randomised clinical trial. Lancet. 2008 Mar 29;371(9618):1085-97. doi: 10.1016/S0140-6736(08)60486-9. PMID 18374841
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Kadam P, Bhalerao S. Sample size calculation. Int J Ayurveda Res. 2010 Jan;1(1):55-7. doi: 10.4103/0974-7788.59946. No abstract available. PMID 20532100
- See also: A clinical case definition of post COVID-19 condition — https://www.who.int/publications/i/item/WHO-2019-nCoV-Post_COVID-19_condition-Clinical_case_definition-2021.1